CLINICAL TRIAL: NCT00256061
Title: Assessment of Electrolyte Values in the Intensive Care Unit:Comparison Between Arterial and Venous Blood Gas Analysis and Formal Laboratory Testing
Status: Withdrawn | Type: Observational
Why Stopped: Due to the publication of significant literature in this area since commencement of the project which has now rendered the project unnecessary.
Sponsor: Melbourne Health (Other)
Other Study IDs: 2002.229
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Electrolyte Values

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study hypothesis is that in critically ill patients there is significant differences between electrolyte levels measured using blood gas analysers and by laboratory techniques, and between levels measured on arterial and venous blood samples.

DETAILED DESCRIPTION:
The sudy hypothesis is that in critically ill patients there is a significant difference between electrolyte levels measured using blood gas analysers and by laboratory techniques, and between levels measured on arterial and venous blood samples.

The study aim is determine the agreement between electrolyte levels measure by formal laboratory serum analysis and point-of-care blood gas analysis.

Also, to determine the agreement between electrolyte levels measured on simultaneous arterial and venous blood samples, using both serum and whole blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years or older admitted to the intensive care unit
2. Patients who have arterial and central venous access insitu for clinical management purposes.
3. Patients who consent to inclusion in the study, or if the patient is not competent, the next of kins' consent.

Exclusion Criteria:

Nil-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-02; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Megan Robertson, MBBS, Principal Investigator — Royal Melbourne Hospital, Intensive Care Unit